CLINICAL TRIAL: NCT06363617
Title: Implementation of the Fatty Liver Index in Primary Care for Patients at Risk of Hepatic Steatosis to Optimize Clinical Control: Randomized Clinical Trial
Brief Title: Implementation of the Fatty Liver Index in Primary Care
Acronym: FLI-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CSAPG-58
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Steatosis; Overweight and Obesity
MeSH Terms: conditions — Fatty Liver; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLI test implementation (Experimental): A training session will be conducted for healthcare professionals on the risks of hepatic steatosis in patients with a body mass index (BMI) equal to or greater than 25. Additionally, professionals will be instructed in the use of the Fatty Liver Index (FLI) tool, validated for assessing the risk of steatosis. This tool will be implemented in the center's computer system, making it accessible via a link for the professionals receiving the intervention.
  Interventions: Other: FLI
- control (No Intervention): This group of healthcare professionals will continue with their usual clinical practice.

INTERVENTIONS:
Other: FLI — Health professionals will use the FLI test in their clinical practice
  Arms: FLI test implementation

SUMMARY:
This trial aims to evaluate the impact on cardiovascular risk control in individuals in risk of being affected by hepatic steatosis through the implementation of a screening test (Fatty Liver Index) in Primary Care. Medical teams in a primary care center will be divided into 2 groups, with one group using the screening test in their clinical practice. The number of interventions on cardiovascular risk occurring in patients attended by each group of medical teams will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 14 years and older.
* Attended at the Basic Care Units (BCU) participating in the Primary Care Center Baix a Mar study.
* Intention to undergo medical follow-up at the study center.
* Body mass index ≥ 25.

Exclusion Criteria:

* Pregnant women
* Alcohol consumption habit (Standard Drink Unit (SDU); one SDU equals 10 grams of alcohol. Risky consumption is considered from 4 SDUs in men and 2 SDUs in women).
* Displaced patients not assigned to the study center.
* Patients classified as Advanced Chronic Care Model or Complex Chronic Patient.
* Participants diagnosed with any of the following pathologies: Chronic liver diseases, including hepatic steatosis; Dementia; Active oncological diseases
* Cognitive or affective pathology that limits the ability to collaborate with lifestyle interventions carried out at the center.
* Patients under the care of endocrinology specialists.
* Participation in another clinical trial involving an experimental intervention during the period of this trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Lifestyle Intervention | Month 6
  Percentage of participants receiving a lifestyle intervention from the start of the study to month 6

SECONDARY OUTCOMES:
Low-density lipoprotein cholesterol | Month 12
  Value of low-density lipoprotein cholesterol (LDL cholesterol) in analyses performed between 6 months and one year post-intervention
Triglycerides | Month 12
  Value of triglycerides in analyses performed between 6 months and one year post-intervention
Gamma-glutamyl transpeptidase | Month 12
  Value of gamma-glutamyl transpeptidase in analyses performed between 6 months and one year post-intervention
Medical and nursing visits | Month 12
  Number of medical and nursing visits in the year following the intervention.
Analytical checks in the first year | Month 12
  Percentage of patients who had not undergone previous analytical checks according to protocol and who undergo analysis in the first year after the start of the study.
Lipid-lowering drugs | Month 12
  Number of prescriptions for lipid-lowering drugs.
Healthcare spending | Month 12
  Analysis of healthcare spending associated with each intervention, using billing data from the center associated with the use of resources by the insured party.
FLI administration | Month 12
  Percentage of patients with body mass index equal or more than 25 who have been administered the FLI

CONTACTS AND LOCATIONS:
Overall Officials: M Carmen Rosas, MD, Principal Investigator — CSAPG
Locations (1):
- Centro de Salud Vilanova i la Geltrú 3 Baix A Mar, Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, CSR
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.